CLINICAL TRIAL: NCT02539628
Title: Adductor Canal Block With Continuous Infusion Versus Intermittent Boluses and Morphine Consumption: A Randomized, Triple-masked, Controlled Study
Brief Title: Adductor Canal Block With Continuous Infusion Versus Intermittent Boluses and Morphine Consumption
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pia Jaeger (Other)
Collaborators: University of California, San Diego (Other); Bispebjerg Hospital (Other); Smiths Medical, ASD, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Pia Jaeger, Sponsor-Investigator, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SM3-PJ-14; 2014-005642-22 (EudraCT Number)
Record Dates: First submitted 2015-03-13; First posted 2015-09-03 (Estimated); Last update posted 2017-04-28 (Actual); Status verified 2017-04

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intermittent bolus (Experimental): ropivacaine 0.2%, 21 ml every 3 hours
  Interventions: Drug: ropivacaine 0.2%
- Continuous infusion (Active Comparator): ropivacaine 0.2%, 7ml/h
  Interventions: Drug: ropivacaine 0.2%

INTERVENTIONS:
Drug: ropivacaine 0.2% — Adductor canal block. Placed immediately postoperative. Intervention stops on POD2 12PM

SUMMARY:
The investigators believe sufficient spread to all nerves within the adductor canal-and thereby sufficient analgesia-can only be obtained by bolus injections and not by continuous infusions via a catheter. The aim of the study is to investigate whether an adductor canal block performed as repeated intermittent boluses provides superior pain relief to continuous infusion. The investigators hypothesize that adductor canal block performed as intermittent boluses via a catheter will reduce morphine consumption and pain as well as enhance ambulation and muscle strength compared with continuous infusion.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for total knee arthroplasty in spinal anesthesia
* Patients who gave their written informed consent to participating in the study after having fully understood the contents of the protocol and restrictions
* American society of anesthesiologists 1-3
* Ability to perform a timed up and go test preoperatively

Exclusion Criteria:

* Patients who cannot cooperate
* Patients who cannot understand or speak Danish.
* Patients with allergy to the medicines used in the study
* Patients with a daily intake of strong opioids (morphine, oxycodone, ketobemidone, methadone, fentanyl) during the last 4 weeks
* Patients suffering from alcohol and/or drug abuse - based on the investigator's assessment
* Rheumatoid arthritis
* BMI > 40
* Neuromuscular pathology in the lower limbs
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2015-03; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Total opioid consumption | 2 days postoperative
  Difference in total opioid consumption (patient controlled analgesia pump and any potential rescue administration) between groups, from end of surgery until 12 pm on postoperative day (POD) 2.

SECONDARY OUTCOMES:
Pains scores during knee flexion as assessed by the Visual analogue scale (VAS) | 2 days postoepratively
  Visual analogue scale (VAS) pain scores (0-100 mm) during 45 degrees active knee flexion analyzed using a linear mixed model with the inclusion of all time points (Day of surgery (DOS): 8 pm, POD 1: 8 am, 12 pm, 8 pm, POD 2: 8 am and 12 pm).
Pain at rest as assessed by the VAS pain scores | 2 days postoperatively
  VAS pain scores (0-100 mm) at rest analyzed using a linear mixed model with the inclusion of all time points (DOS: 8 pm, POD 1: 8 am, 12 pm, 8 pm, POD 2: 8 am and 12 pm).
Pain during the Timed Up and Go test as assessed by the VAS | 1 and 2 days postoperatively
  Worst pain (VAS, 0-100 mm) during the Timed Up and Go test at 12 pm on POD 1 and 2.
Quadriceps strength assessed as maximum voluntary isometric contraction in percentage of preoperative baseline values at 12 pm on POD 1 and 2 | 1 and 2 days postoperatively
  Quadriceps strength assessed as maximum voluntary isometric contraction in percentage of preoperative baseline values at 12 pm on POD 1 and 2.
Timed Up and Go test | 1 and 2 days postoperatively
  Time (seconds) to perform the Timed Up and Go test at 12 pm on POD 1 and 2.
Number of patients able to perform the Timed Up and Go test | 1 and 2 days postoperatively
  Number of patients able to perform the Timed Up and Go test at 12 pm on POD 1 and 2.
6 min walk test | 1 and 2 days postoperativley
  Distance ambulated (m) during the 6 min walk test performed at 12 pm on POD 1 and 2.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anaesthesia-Surgery-Intensive Care, Gentofte Hospital, Gentofte Municipality, Hellerup, Denmark

REFERENCES:
- [Derived] Jaeger P, Baggesgaard J, Sorensen JK, Ilfeld BM, Gottschau B, Graungaard B, Dahl JB, Odgaard A, Grevstad U. Adductor Canal Block With Continuous Infusion Versus Intermittent Boluses and Morphine Consumption: A Randomized, Blinded, Controlled Clinical Trial. Anesth Analg. 2018 Jun;126(6):2069-2077. doi: 10.1213/ANE.0000000000002747. PMID 29293181